CLINICAL TRIAL: NCT04416282
Title: Efficacy of Early Terlipressin Plus Albumin Therapy in Comparison to Standard Treatment for HRS-AKI in Acute-on-chronic Liver Failure- A Randomized Open Label Study.
Brief Title: Efficacy of Early Terlipressin Plus Albumin Therapy in Comparison to Standard Treatment for HRS-AKI in Acute-on-chronic Liver Failure.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ACLF-04
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Acute-On-Chronic Liver Failure; Hepatorenal Syndrome; Acute Kidney Injury
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatorenal Syndrome; Acute Kidney Injury | interventions — Terlipressin; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terlipressin + Albumin (Experimental): Injection terlipressin 2 mg/24 hours infusion + i/v albumin 1g/Kg/day
  Interventions: Drug: Terlipressin; Biological: Albumin
- Albumin (Active Comparator): i/v albumin 1g/Kg/day for next 36 hours f/b inj terlipressin 2mg/24 hours
  Interventions: Biological: Albumin

INTERVENTIONS:
Drug: Terlipressin — Injection terlipressin 2 mg/24 hours infusion
  Arms: Terlipressin + Albumin
Biological: Albumin — i/v albumin 1g/Kg/day

SUMMARY:
Acute on chronic liver failure (ACLF) is a distinct entity where, because of severe acute hepatic injury, a rapid loss of liver function develops in a patient with previous chronic liver disease(4). These patients have severe hepatic dysfunction, and outcome is defined by functional hepatic reserve and extent of extra-hepatic organ failures(5). Renal failure is a frequent extra-hepatic organ failure, and its presence is an independent prognostic marker for mortality(12). The pathophysiological basis of renal dysfunction in patients with ACLF is different compared to those with decompensated cirrhosis (DC)(6). Systemic inflammation is the hallmark of ACLF, characterized by a cytokine storm wherein there is an increase in both pro- and anti-inflammatory cytokines, such as interleukin (IL)-6, IL-8, IL-1β, and IL-10, leading to circulatory dysfunction and organ failure(3). These patients therefore have a higher incidence and progression of acute kidney injury (AKI). Diagnosis of HRS-AKI in ACLF currently requires 48 h of volume repletion with albumin and diuretic withdrawal. Therefore waiting for 48 hours to start treatment with terlipressin can be associated with worsening of AKI stage, worsening of ACLF stage and thereby suboptimal treatment response and high mortality despite treatment response. Therefore early initiation of terlipressin as continuous infusion after volume repletion with IV albumin in ACLF-AKI is safe and prevents AKI progression by splanchnic vasoconstriction and improved renal perfusion.

DETAILED DESCRIPTION:
Aim To compare the effect of Early initiation of Terlipressin (ET arm) to albumin at 12 hour in ACLF patients with non-volume responsive AKI versus standard Terlipressin (ST arm) at 48 hours.

Primary Objective Efficacy of early terlipressin infusion in comparison to Standard treatment for resolution of AKI at day 7.

Secondary Objectives

* Full and partial AKI response at 48 and 72 h and 96 hours
* Mortality at Day 28, Day 90
* Baseline organ failure(s), MELD, CLIF-SOFA score and ACLF score
* New onset organ failures
* Urine Output
* Progression or resolution of OFs at day 7
* Change in MELD, CLIF-SOFA score and ACLF score at day 7
* Change in NGAL, FENa, FE-Urea at day 7
* Treatment related adverse effects and their grades

Methodology:

Study population:

All patients admitted to the Institute of Liver and Biliary Sciences (ILBS) with ACLF with AKI- HRS will be evaluated for inclusion. ACLF will be defined by the APASL criteria.

Study Design A prospective, randomized, single center open label study

Study Period:Two year

Intervention & monitoring:

Clinical Protocol An informed consent will be taken from ACLF patients with AKI within 24-hours of admission. No alteration in the treatment or investigative procedures of the included patients will be done. All included patients will be followed from admission till death or discharge. All discharged patients will then be followed till 30-days.

Preliminary work up

At admission:

(A) Complete history and physical examination

* Recent Diuretics use
* Loose stools
* Recurrent vomiting
* Fever, signs of sepsis (SIRS)
* H/s/o LRTI, SSTI, SBP
* Recent contrast use (< 7 days)
* Use of nephrotoxins including NSAIDs
* Prior renal dysfunction, known CKD, HD
* History of HTN, Diabetes
* History of renal stones
* History s/o hypotensive episodes (shock)

Pre-randomization interventions:

(B) Intervention during 0-12 hours (Before randomization) -

* Withdrawal of diuretics
* Withdrawal of lactulose (in patients with loose stools)
* Urine output monitoring (catheterize and monitor hourly or 12 h cumulative)
* 2 hourly MAP, Pulse rate
* Empirical IV antibiotics to be given in case of suspected/proven sepsis (Avoid nephrotoxic drugs e.g Amikacin, Colistin, Amphotericin etc as possible)
* IV hydration with albumin at 12 hours preferably 40 g (20 %) + 500 ml crystalloids)

Labs and follow-up:

* Baseline (at admission) - Blood : KFT, LFT, CBC, INR, Blood c/s, pro-BNP Imaging : USG abdomen, USG KUB, Renal doppler, C-X-ray, 2D ECHO Urine : Urine R/E and cultures, Urine Na, Urea, NGAL, Creatinine, FENa, FE Urea A/F analysis - for SBP
* At 12 hours (Before randomization) - Blood - KFT
* At D1, D2, D3, D5, D7, D14, D28 post randomization Blood : KFT Urine : Urine Na, Urea, NGAL, Creatinine, FENa, FE Urea (At Day 3 and 7) Imaging : Renal doppler (Day 3)

Clinical evaluation:

* Etiology of cirrhosis (Baseline)
* Severity of liver disease (Baseline, D3, D7) MELD score, CLIF-SOFA score, MELD-Na score, AARC score
* Stage of ACLF (Baseline,D3, D7) AARC grade, CLIF ACLF grade
* Complications / Organ failures (Baseline,D3, D7) HE, Bleed, AKI stage, SBP, Infection (specify site and severity) Respiratory and circulatory failure

Follow up duration Duration of admission till discharge or death will be noted. Patients will be followed up to 28-days for re-admission(s) and survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years
2. ACLF as per APASL criteria
3. AKI at admission as defined by ICA-AKI criteria
4. AKI stage 2/3 at 12 hour of admission

Exclusion Criteria:

-

At Admission:

* Age <18 years
* Patients on renal replacement therapy (RRT)
* Post renal or liver transplantation
* History of CAD, ischemic cardiomyopathy, PVD, ventricular arrhythmia
* Decompensated cirrhosis not fulfilling ACLF criteria
* Cirrhotics with AKI managed as outpatients
* Grade III/IV HE or Shock requiring inotropes or patients on mechanical ventilator at time of randomization
* In-hospital new AKI
* Active urinary sediments - 2+ albumin or above, dysmorphic RBCs
* Known CKD, obstructive uropathy
* Lack of informed consent
* Prior intolerance or S/E to Terlipressin or albumin

At 12 Hour before randomization:

• Regression of AKI (>0.3 mg/dl) above baseline after IV albumin (20% 40 gm) + IV Crystalloids 500 ml therapy for 12 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Acute Kidney Injury reversal by day 7 in both groups | Day 7

SECONDARY OUTCOMES:
Mortality in both groups | Day 28
Mortality in both groups | Day 90
Progression or resolution of Organ failures | Day 90
Adverse Events in both groups | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided